CLINICAL TRIAL: NCT07098065
Title: Effectiveness of Health Warnings and Counseling at Primary Health Care Centers for Smoking Cessation and NCD Prevention: Study Protocol for a Cluster Randomized Controlled Trial in Bangladesh and Pakistan
Brief Title: Health Warnings and Counseling for Smoking Cessation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hitotsubashi University (Other)
Collaborators: Global Public Health Research Foundation (Other)
Responsible Party: Principal Investigator, Md. Mizanur Rahman, PhD, Associate Professor, Hitotsubashi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GHW Trial for smokers
Record Dates: First submitted 2025-07-23; First posted 2025-08-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Tobacco Cessation; Health Warning Label; Hypertension; Non Communicable Chronic Diseases
Keywords: Tobacco cessation; Graphic health warnings (GHWs); Non-communicable diseases (NCDs); Cluster randomized controlled trial (RCT); Pharmacist-led counseling
MeSH Terms: conditions — Tobacco Use Cessation; Hypertension; Noncommunicable Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GHW-only intervention (Experimental): This group will receive only graphical health warnings (GHWs) featuring images proposed by the Bangladesh Tobacco Control Cell, explicitly illustrating smoking-related harms, such as mouth diseases, damaged teeth and gums, lung diseases and cancer, heart diseases and cardiovascular damage, and throat and oral cancer. Additionally, these warnings will clearly highlight the benefits of quitting smoking-including improved overall health, reduced disease risks, financial savings, and enhanced quality of life-as well as practical cessation techniques. Participants will receive these GHW materials at baseline and again at the six-month follow-up to reinforce these critical health messages; however, this intervention group will not receive any counselling services. Monthly SMS reminders will also be sent to participants, prompting them to review the GHW leaflet and reinforcing the negative health impacts of smoking and the benefits of quitting.
  Interventions: Behavioral: Graphical health warnings
- GHW plus pharmacist-led counselling (Experimental): Participants in this group will receive graphical health warnings (GHWs) featuring Bangladesh Tobacco Control Cell-approved images clearly depicting smoking-related harms (e.g., mouth diseases, damaged teeth and gums, lung cancer, heart disease, and oral cancer). Additionally, they will receive personalized counselling from community pharmacists, focused on the specific health and financial benefits of quitting, practical cessation techniques, strategies for overcoming barriers, and relapse prevention. This combined intervention will be provided at baseline and reinforced at a six-month follow-up. Monthly SMS reminders will also be sent, reinforcing key messages on the harmful effects of smoking and benefits of cessation.
  Interventions: Behavioral: Graphical health warnings plus pharmacist-led counselling
- Standard care control (Active Comparator): Participants in this group will receive only routine pharmacy services based on standard pharmacy practice guidelines applicable in each country. They will not receive any additional graphical health warnings or counselling interventions. Outcomes will be assessed at baseline, 6 months, and 12 months, consistent with the intervention groups.
  Interventions: Other: Routine pharmacy services (no intervention)

INTERVENTIONS:
Behavioral: Graphical health warnings — This group will receive only graphical health warnings (GHWs) featuring images proposed by the Bangladesh Tobacco Control Cell, explicitly illustrating smoking-related harms, such as mouth diseases, damaged teeth and gums, lung diseases and cancer, heart diseases and cardiovascular damage, and throat and oral cancer. Additionally, these warnings will clearly highlight the benefits of quitting smoking-including improved overall health, reduced disease risks, financial savings, and enhanced quality of life-as well as practical cessation techniques. Participants will receive these GHW materials at baseline and again at the six-month follow-up to reinforce these critical health messages; however, this intervention group will not receive any counselling services. Monthly SMS reminders will also be sent to participants, prompting them to review the GHW leaflet and reinforcing the negative health impacts of smoking and the benefits of quitting.
  Arms: GHW-only intervention
Behavioral: Graphical health warnings plus pharmacist-led counselling — Participants in this group will receive graphical health warnings (GHWs) featuring Bangladesh Tobacco Control Cell-approved images clearly depicting smoking-related harms (e.g., mouth diseases, damaged teeth and gums, lung cancer, heart disease, and oral cancer). Additionally, they will receive personalized counselling from community pharmacists, focused on the specific health and financial benefits of quitting, practical cessation techniques, strategies for overcoming barriers, and relapse prevention. This combined intervention will be provided at baseline and reinforced at a six-month follow-up. Monthly SMS reminders will also be sent, reinforcing key messages on the harmful effects of smoking and benefits of cessation.
  Arms: GHW plus pharmacist-led counselling
Other: Routine pharmacy services (no intervention) — Participants in this group will receive only routine pharmacy services based on standard pharmacy practice guidelines applicable in each country. They will not receive any additional graphical health warnings or counselling interventions. Outcomes will be assessed at baseline, 6 months, and 12 months, consistent with the intervention groups.
  Arms: Standard care control

SUMMARY:
Tobacco use remains persistently high across South Asia, despite numerous public health efforts, and continues to significantly contribute to the burden of non-communicable diseases (NCDs) such as cardiovascular disease, hypertension, diabetes, and stroke. Community pharmacists-widely accessible and trusted within their communities-are an underutilized resource for delivering public health interventions. Graphic health warnings (GHWs), recommended by the World Health Organization (WHO), have been shown to promote smoking cessation, but are rarely paired with personalized counseling by healthcare providers.

This study aims to evaluate both the effectiveness and cost-effectiveness of integrating GHWs with pharmacist-led personalized counseling at primary healthcare pharmacies in Bangladesh and Pakistan. A cluster randomized controlled trial (RCT) will be conducted, enrolling 5,052 adult participants in each country from community pharmacies. Participants will be randomly assigned to one of three groups: (1) GHW-only intervention, (2) combined GHW and pharmacist-led counseling, or (3) standard care (control).

The intervention includes twice-yearly counseling sessions-delivered both in-person and digitally-supported by educational booklets and leaflets. Primary outcomes are smoking cessation rates and blood pressure reduction. Secondary outcomes include improved hypertension and diabetes management, medication adherence, lifestyle modification, reduced hospitalizations and mortality, and incremental cost-effectiveness. Bayesian statistical models will be used to assess efficacy, and economic evaluations will determine the cost-effectiveness of the interventions. The findings aim to inform scalable public health strategies for tobacco control and NCD prevention in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older
* Regular pharmacy visitors who currently smoke or have medically diagnosed hypertension without organ damage
* Permanent resident of the study area,
* Access to mobile phone
* Able to operate smartphone or tablet.

Exclusion Criteria:

* Without pregnancy and lactation
* Without cognitive or psychiatric conditions,
* Without severe medical conditions,
* Participation in other studies, and inability to consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5052 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Verified smoking cessation rates | Baseline, 6 months, and 12 months post-intervention.
  Percentage of participants who report smoking cessation
Change in Systolic Blood Pressure (SBP) | Baseline, 6 months, and 12 months.
  Mean change in systolic blood pressure (mmHg) from baseline to 6 and 12 months. Changes in Blood pressure in the target intervention group (Whose SBP<140 mmHg and DBP<90 mmHg were in the baseline) Changes in SBP and DBP of the patients at baseline, at 12 months and 18 months post-intervention.
  Changes in Blood pressure in the target intervention group (Whose SBP<140 mmHg and DBP<90 mmHg were in the baseline)
Change in Diastolic Blood Pressure (DBP) | Baseline, 6 months, and 12 months.
  Mean change in diastolic blood pressure (mmHg) from baseline to 6 and 12 months.
Change in Quality-Adjusted Life Years (QALYs) | Baseline, 6 months, and 12 months.
  Incremental QALYs gained from baseline to 12 months, based on health utility measures (e.g., EQ-5D).
Improvement in Knowledge About Smoking Harms | Baseline, 6 months, and 12 months.
  Percentage increase in correct responses to questions on the health effects of smoking.

SECONDARY OUTCOMES:
Improved Hypertension Management | 6 and 12 months.
  Proportion of hypertensive participants achieving BP <140/90 mmHg or reporting medication adherence.
Improved Diabetes Management | 6 and 12 months.
  Proportion of participants with diabetes reporting glucose monitoring, medication adherence, or controlled HbA1c (if available).
Hospital Admissions | 6 and 12 months.
  Number of participants reporting hospital admission related to NCDs (e.g., hypertension, stroke, cardiac events).
All-Cause Mortality | Up to 12 months.
  Number of deaths (any cause) among enrolled participants during the study period.
Increase in Physical Activity | 6 and 12 months.
  Increase in days per week with at least 30 minutes of moderate activity.
Incremental Cost-Effectiveness Ratio | At 12 months.
  Cost per QALY gained comparing intervention arms to control.
Image-Based Biomarker Assessment (Exploratory Secondary Outcome) | Time Frame: Baseline and 12 months.
  Quantitative features extracted from facial photographs, eye photographs, and chest X-rays will be analyzed to examine associations with smoking exposure, blood pressure, and cardiometabolic risk markers.

CONTACTS AND LOCATIONS:
Overall Officials: Md. Mizanur Rahman, Principal Investigator — Hitotsubashi University
Locations (1):
- Global Public Health Research Foundation, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No